CLINICAL TRIAL: NCT06455137
Title: Epidural Electrical Stimulation for Spinal Cord Injury Patients and Corticospinal Motor Circuit Improvement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB112-067-A
Record Dates: First submitted 2024-06-07; First posted 2024-06-12 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Epidural Stimulator (Experimental): Participants will have a 16-electrode epidural array implanted in the C4-C7 and T11-L2 areas of the spinal cord. Following a 2 weeks recovery period, patients will engage in a structured training of physical rehabilitation and electrical stimulation.
  Interventions: Device: Epidural Stimulator

INTERVENTIONS:
Device: Epidural Stimulator — Participants will have a 16-electrode epidural array implanted in the C4-C7 and T11-L2 areas of the spinal cord. Following a 2 weeks recovery period, patients will engage in a structured training of physical rehabilitation and electrical stimulation.

SUMMARY:
The study aims to examine the plausible interventional mechanisms underlying the effects of epidural spinal cord stimulation.

DETAILED DESCRIPTION:
The purpose of this study is for the treatment of spinal cord injury (SCI) paralysis patients use the signal by electrophysiological analysis of epidural spinal cord stimulation (SCS) settings that promote limbs activity so that SCI patients can restore motor ability under multiple sensory stimuli and multimodal electrical stimulation rehabilitation. The investigators hope to establish an atresia nerve regulation strategy and observe that the original blocked neural circuits can improve nerve plasticity by SCS. Even can establish new connections through residual nerves and allow SCI patients to rebuild neural circuits without SCS to restore limbs mobility and improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* SCI ASIA: A, B, C,D
* Between 20 and 70 year of age
* >1 year post SCI
* Complete or incomplete spinal cord injury.
* Expected will undergo spinal cord stimulation surgery.
* Continued rehabilitation after surgery for spinal cord injury.
* Able to comply with procedures and follow up.
* Stable medical condition without cardiopulmonary disease or dysautonomia that would - contraindicate participation in lower extremity rehabilitation or testing activities

Exclusion Criteria:

* Have significant cognitive impairment (MMSE<24).
* Had a mental illness within one year or been treated in the past.
* Have Major depressive disorder.
* Active cancer diagnosis.
* Painful musculoskeletal dysfunction, unhealed fracture, contracture, pressure sore, or urinary tract infection that might interfere with stand or step training.
* Cardiovascular or musculoskeletal disease or injury that would prevent full participation in physical therapy intervention.
* Unable to read and/or comprehend the consent form.
* Have concerns about this trial and do not sign consent.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Electroencephalography and Electromyography | To measure assessing change between pre-implant and every 3 months until 24 months.
  To measure activity in the brain
Electromyographic analysis | To measure assessing change between pre-implant and every 3 months until 24 months.
  Average of 5-repetitive EMG activity for each superficial component of muscles from a five-second ramp contraction to the end of a ten-second rest
Single transcranial magnetic stimulation | To measure assessing change between pre-implant and every 3 months until 24 months.
  To evaluate the function of corticospinal tract nerve conduction
Motion Analysis | To measure assessing change between pre-implant and every 3 months until 24 months.
  To evaluate the angles that can be achieved at each joint of the upper limbs
Functional Test | To measure assessing change between pre-implant and every 3 months until 24 months.
  To evaluate gait for subjects who can walk by assistive device or independently

SECONDARY OUTCOMES:
American Spinal Injury Association (ASIA-2019) Impairment Scale | To measure assessing change between pre-implant and every 3 months until 24 months.
  To measure and record disease history
  In simpler terms, it's a 5-point scale that categorizes individuals from "A" (complete spinal cord injury) to "E" (normal sensory and motor function), with each letter representing a different level of injury severity:
  A: Complete spinal cord injury. B: Sensory incomplete injury. C: Motor incomplete injury. D: Motor incomplete injury. E: Normal sensory and motor function.
Modified Ashworth scale | To measure assessing change between pre-implant and every 3 months until 24 months.
  To measure the increase of muscle tone,it uses a 6-point system. Scores range from 0 to 4. Lower scores indicate normal muscle tone, while higher scores indicate spasticity or increased resistance to passive movement.
Barthel Index | To measure assessing change between pre-implant and every 3 months until 24 months.
  To measure performance in activities of daily living
World Health Organization Quality of Life Brief Version | To measure assessing change between pre-implant and every 3 months until 24 months.
  A brief version scale of World Health Organization Quality-of-Life scale
Spinal Cord Independence Measure | To measure assessing change between pre-implant and every 3 months until 24 months.
  To measure performance in activities of daily living and mobility
Box and Block Test | To measure assessing change between pre-implant and every 3 months until 24 months.
  To measure unilateral gross manual dexterity.
Action Research Arm Test Scoring Sheet | To measure assessing change between pre-implant and every 3 months until 24 months.
  To measures upper limb function by scoring the ability to complete functional tasks.
Berg Balance Scale | To measure assessing change between pre-implant and every 3 months until 24 months.
  To measure balance and the risk of falls,it's a list of 14 things to rate, where each thing has a scale from 0 to 4. Zero means the lowest function, while four means the highest function.
Walking Index for Spinal Cord Injury II (WISCI II- March 2005) | To measure assessing change between pre-implant and every 3 months until 24 months.
  To measure walking ability for spinal cord injury.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Tzung Tsai, M.D., Ph.D., Principal Investigator — Hualien Tzu Chi General Hospital
Locations (1):
- Buddhist Tzu Chi Medical Foundation Hualien Tzu Chi Hospital, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No